CLINICAL TRIAL: NCT01369160
Title: Curative vs Disease-Modifying Therapies in Children With Severe Sickle Cell Disease: A Pilot, Cross-Sectional Study
Brief Title: Curative Versus Disease-Modifying Therapies in Children With Severe Sickle Cell Disease
Acronym: SCD_Cross
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ann E. Haight, Assistant Professor, Emory University
Other Study IDs: 261-2005
Record Dates: First submitted 2009-04-22; First posted 2011-06-08 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Chronic Transfusion
  Interventions: Behavioral: Quality of Life measures
- 2: hydroxyurea
  Interventions: Behavioral: Quality of Life measures
- 3: matched sibling donor stem cell transplantation (MSD-SCT)
  Interventions: Behavioral: Quality of Life measures
- 4: standard comprehensive care (SCC, control)
  Interventions: Behavioral: Quality of Life measures

INTERVENTIONS:
Behavioral: Quality of Life measures — measuring QOL with different therapies

SUMMARY:
The research proposed is a pilot study of pediatric and adolescent/young adult patients who have received the curative intervention (MSD-SCT), disease-modifying interventions (HU or CT) or SCC (control), with respect to three clinically important outcomes: quality-of-life (QOL), neurocognitive function, and reproductive potential. Comparable cohorts will be identified for each of the groups, drawing from patients treated by the SCD program of Children's Healthcare of Atlanta (CHOA). QOL measures and neuropsychiatric testing and will be administered. Reproductive endocrine function markers (laboratory studies and pubertal staging), will be collected and analyzed. A tracking system of such patients will also be developed, gathering available retrospective data and setting up a mechanism for collection of new data.

DETAILED DESCRIPTION:
sickle cell disease (SCD), but a significant proportion experience clinically severe disease requiring more aggressive intervention. Widely applicable curative therapy with a favorable toxicity profile remains elusive for such patients.

Three distinct intervention strategies are currently available for children with severe sickle cell disease (SCD): oral hydroxyurea (HU), chronic blood transfusions (CT), and allogeneic hematopoietic stem cell transplantation (SCT) from an HLA-matched sibling donor (MSD). Each intervention has distinct advantages and disadvantages. Many patients do not receive specific intervention, and continue standard comprehensive care (SCC).

Though indications for these therapies overlap, to date there are no comparative outcomes data, leaving families and physicians without adequate information upon which to base therapeutic decisions. The gold standard for obtaining such data would be a randomized, prospective study comparing each intervention, though this may or may not be feasible to conduct. Before such a trial is considered, a large cross-sectional trial should be conducted to establish comparisons among the four therapeutic groups (HU, SCT, CT, SCC) with respect to the outcomes that clinicians and families deem most important.

The research proposed is a pilot study of pediatric and adolescent/young adult patients who have received the curative intervention (MSD-SCT), disease-modifying interventions (HU or CT) or SCC (control), with respect to three clinically important outcomes: quality-of-life (QOL), neurocognitive function, and reproductive potential. Comparable cohorts will be identified for each of the groups, drawing from patients treated by the SCD program of Children's Healthcare of Atlanta (CHOA). QOL measures and neuropsychiatric testing and will be administered. Reproductive endocrine function markers (laboratory studies and pubertal staging), will be collected and analyzed. A tracking system of such patients will also be developed, gathering available retrospective data and setting up a mechanism for collection of new data.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 3 years of age
* Homozygous hemoglobin S (HbSS)
* Severe disease, defined as having one or more of the following:
* recurrent (2 or more episodes per year) acute chest syndrome (ACS),
* frequent (3 or more episodes per year) vaso-occlusive pain events, defined as episode lasting 4 hours and requiring hospitalization or outpatient treatment with parenteral narcotics
* Any combination of 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years.
* any stroke, defined as central nervous system (CNS) event lasting longer than 24 hours, plus objective imaging evidence of CNS vasculopathy, with or without residual neurologic findings
* At least one year has elapsed since start of therapy for severe disease (CT, HU, MSD-BMT or SCC).

Exclusion Criteria:

* Inadequate medical records to support eligibility criteria
* Patients less than 1 year from start of therapy (CT, HU, MSD-BMT or SCC).

Ages: 3 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
quality of life | 5 years after last patient enrolled
neuropsychiatric testing | 1 year after last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haight, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia